CLINICAL TRIAL: NCT06100042
Title: Multicentre, Prospective, Non-interventional Study Monitoring Therapy Pathways of Asthma Patients Treated With an Extrafine ICS/LABA/LAMA Single-inhaler Triple Therapy in a Real-world Setting and Characterizing the Effects on Health-related Outcomes
Brief Title: Observational Study on Therapy Pathways of Asthamics Treated With ICS/LABA/LAMA Therapy in a Real-world Setting
Acronym: TRIMAXIMIZE
Status: Active, not recruiting | Type: Observational
Sponsor: Chiesi Italia (Industry)
Collaborators: Gesellschaft für Therapieforschung mbH (Industry)
Responsible Party: Sponsor
Organization: Chiesi Farmaceutici S.p.A. (Industry)
Other Study IDs: CHIT-2301; NIS 005 Pn (Other: International study code)
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Asthma
Keywords: Asthma; Triple Therapy; Beclomethasone; Formoterol; Glycopyrronium; Real-world; Single-Inhaler; Quality of life; Control of asthma; Adherence
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Asthma patients: Adult patients with a diagnosis of moderate to severe asthma treated with BDP/FF/G medium strength or high strength as per clinical practice.
  Interventions: Drug: BDP/FF/G

INTERVENTIONS:
Drug: BDP/FF/G — BDP/FF/G is an extrafine single inhaler triple therapy available in two dosage strengths:
  * Medium strength (MS) containing 100 µg of beclomethasone dipropionate, 6 µg of formoterol fumarate dihydrate and 10 µg of glycopyrronium (as 12.5 µg glycopyrronium bromide);
  * High strength (HS) containing 200 µg of beclomethasone dipropionate, 6 µg of formoterol fumarate dihydrate and 10 µg of glycopyrronium (as 12.5 µg glycopyrronium bromide).
  Other Names: Trimbow

SUMMARY:
TriMaximize is a non-interventional study aimed to collect prospective data from asthmatic patients under routine care, for whom their treating physician has decided to prescribe BDP/FF/G (beclomethasone/formoterol/glycopyrronium).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age;
* Patients with confirmed leading diagnosis of asthma with or without concomitant COPD;
* Physician decision to start fixed triple therapy with ICS/LABA/LAMA (BDP/FF/G) MS or HS according to its current authorised indication and current reimbursement conditions within the Italian National Health System. The treatment decision must be made independently from participation in this study and may have started within the previous 4 weeks (maximum);
* Patients willing and able to sign an informed consent for use of their pseudonymised clinical data within the present non-interventional study.

Exclusion Criteria:

* Participation in an interventional clinical trial within 30 days prior to enrolment into the present non-interventional study or planned enrolment in an interventional clinical trial during the observational period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a diagnosis of moderate to severe asthma treated with BDP/FF/G as per clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient demographics | 12 months

SECONDARY OUTCOMES:
Assessment of asthma control using Asthma Control Test (ACT) | 12 months
  Change from baseline in ACT scores. The ACT is a self-report questionnaire with scores ranging from 5-25 (higher is better). Scores of 20-25 are classified as well-controlled; 16-19 as not well-controlled; and 5-15 as very poorly controlled asthma. The minimum clinically important difference is considered to be 3 point.
Assessment of quality of life using Mini Asthma Quality of Life Questionnaire (Mini AQLQ) | 12 months
  Change from baseline in MiniAQLQ scores. The MiniAQLQ is a disease specific questionnaire that consists of 15 asthma-related questions.
  Participants respond to each question on a 7-point scale (1=severe impairment, 7=no impairment), where higher scores indicated better quality of life. A change in the score greater than 0.5 can be considered clinically important.
Assessment of adherence to treatment using 12-item Test of Adherence to Inhalers (TAI-12) | 12 months
  Change from baseline in TAI-12 score. The 12-item TAI comprises a patient domain (10 items) and a healthcare professional domain (2 items).
  Each item ranges from 1 (lowest adherence) to 5 (highest adherence) points. The patient domain score ranges from 10 to 50. Adherence is rated as good (score = 50), intermediate (score = 46-49).
Incidence of asthma exacerbations | 12 months
  Number of exacerbations
Asthma exacerbations | 12 months
  Occurrence of asthma exacerbations
Adverse events | 12 months
  Number of AEs
Adverse drug reactions to BDP/FF/G | 12 months
  Number of ADRs

CONTACTS AND LOCATIONS:
Locations (1):
- U.O. Clinica Psichiatrica e SPDC. Ospedale Policlinico S. Martino - IRCCS, Genova, Genoa, Italy

IPD SHARING:
Plan to Share IPD: No